CLINICAL TRIAL: NCT03576170
Title: Investigate the Efficacy and Effectiveness of Aromatherapy for the Management of Behavioral and Psychological Symptoms of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor and Head Department of Rehabilitation Science, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P17-0203-1
Record Dates: First submitted 2018-06-08; First posted 2018-07-03 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aromatherapy-scent (Active Comparator)
  Interventions: Other: aromatherapy
- aromatherapy-touch (Active Comparator)
  Interventions: Other: aromatherapy
- wait-list control (No Intervention)

INTERVENTIONS:
Other: aromatherapy — aromatherapy by inhalation and/or therapeutic massage
  Arms: aromatherapy-scent; aromatherapy-touch

SUMMARY:
In recent decades, following an increased longevity in Hong Kong, there is a drastic increase in the prevalence chronic conditions, including dementia. Behavioral and psychological symptoms of dementia (BDSP) seem to be the main reasons of suffering for many older adults. This condition does not only pose a burden to the whole family but also the healthcare system.

While conventional treatment of BPSD using pharmacotherapy and non-pharmacological treatments has been effective for managing symptoms, owing to the adverse side effects caused by anti-psychotic drugs and the short effective period incurred by non-pharmacological interventions, development of alternative and non-pharmacological approaches for the management of behavioral disturbances and pain is of urgent need. Research has shown that aromatherapy (both administered through inhalation and therapeutic massage) has been effective in reducing behavioral disturbances of dementia patients. These findings support the premise that aromatherapy and the investigators hope to provide further evidence to support the use of aromatherapy as an evidence-based mainstream intervention for reducing behavioral and psychological symptoms of dementia (BPSD).

Whilst there is sufficient evidence to support the effectiveness of aromatherapy, few studies compared the effectiveness of the use of aromatherapy by inhalation and/or therapeutic massage. The investigators aim to address the above research gaps on the clinical application of aromatherapy on BPSD, with a focus on comparing the differential effectiveness between administration by inhalation and administration by therapeutic massage. The proposed research aims to (1) test the efficacy and effectiveness of aromatherapy on the symptom management of BPSD in older adults; (2) compare the effects of aromatherapy-scent (i.e., inhalation) and aromatherapy-touch (i.e., therapeutic massage) in older adults with BPSD. This study also explores the benefits of aromatherapy on cognitive functioning, functional performance and social engagement as secondary outcomes.

A randomized, controlled, and single blinded trial is proposed. 120 older adults with BPSD will be randomly assigned to aroma inhalation (intervention), aroma-touch or wait-list (control) treatments. The primary outcomes measured are a caregiver-rated inventory of agitated behaviors and abnormalities of mood and psychotic phenomenal, cognitive functioning, functional performance and social engagement (secondary outcome) will be assessed three time points the study hypotheses are supported, the findings will provide empirical support for a treatment option that could improve psychological well-being and also improve cognitive functioning, functional performance, and social engagement of older adults.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* have a CMMSE score below 18 if illiterate, 19 if they have 1-2 years of education, and 20 if they had more than 2 years of education
* reported to have BPSD;
* willing to participate in the research, with informed consent signed by their guardian or carer.

Exclusion Criteria:

* allergic to essential oils
* refused to give consent
* over-sensitive to tactile stimulation
* have a history of kidney and liver disease
* have ever had an epileptic seizure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Chinese Version of the Cohen- Mansfield Agitation Inventory (CMAI) | baseline, 2-months after intervention and after the completion of the intervention in four months
  It is a care-giver rated inventory to assess agitation in elderly persons and records the frequency of occurrence of BDSP at different period of time and thus can be used for assessing the changes among three times points (baseline, 2-months after intervention and after the completion of the intervention) in four months. It includes descriptions of 29 agitated behaviors, and each is rated on a 7-point scale of frequency. The total scores range from 29 points to 203 points, a higher score of CMAI indicates more frequent agitation behaviors.
Chinese Version of the Neuropsychiatric Inventory (NPI) | baseline, 2-months after intervention and after the completion of the intervention in four months
  It is used to assess the changes of the abnormalities of mood and psychotic phenomena among three times points (baseline, 2-months after intervention and after the completion of the intervention) in four months. If the response to the domain question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations on them (i.e. Caregiver Distress) using a 5-point scale. The NPI-Q provides symptom Severity and Distress ratings for each symptom), and total Severity and Distress scores reflecting the sum of individual domain scores ranging from 0 to 36 and ranging from 0 to 60 respectively.

SECONDARY OUTCOMES:
Cantonese Version of the Mini-mental State Examination (CMMSE) | baseline, 2-months after intervention and after the completion of the intervention in four months
  Cantonese Version of Mini-mental State Examination (MMSE) is a brief 30-point questionnaire used to assess the change of the cognitive functions among three time points (baseline, 2-months after intervention and after the completion of the intervention) in four months. The range of the score is from 0 point to 30 points, which a lower score indicates the worse cognitive functions.
Chinese Version of the Barthel Index-100 | baseline, 2-months after intervention and after the completion of the intervention in four months
  Chinese Version of the Barthel Index-100 is used to measure the change of the performance in activities of daily living (ADL) among three time points (baseline, 2-months after intervention and after the completion of the intervention) in four months. Scores range from 0 to 100, with higher scores indicating greater independence.
  of performance in basic activities of daily living (BADL) which is sensitive to either decline or improvement on the functional level of the elderly
Chinese Version of the Index of Social Engagement(ISE) | baseline, 2-months after intervention and after the completion of the intervention in four months
  The change of the social engagement among three time points (baseline, 2-months after intervention and after the completion of the intervention) in four months will be measured using the 6-item index of social engagement (ISE). Total scores on the ISE can range from 0 to 6, with a higher score indicating a higher level of social engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechinic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No